CLINICAL TRIAL: NCT04160403
Title: The Factors as Socioeconomic Status and Child Characteristics That May Impact on the Progress of Development After Physical Therapy Interventions in Children With Spastic Cerebral Palsy
Brief Title: The Socioeconomic Status and Child Characteristics on the Physical Therapy Outcome in Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeinab Hussein (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Zeinab Hussein, professor, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P.T.REC/012/001761
Record Dates: First submitted 2019-11-09; First posted 2019-11-13 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-11

CONDITIONS: C10.228.140.140.254
Keywords: Cerebral palsy, spastic, motor function, socioeconomic status, progress, physical therapy
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: prospective cohort study
Masking Description: the data about socioeconomic status did not be announced
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- factors ( SES,age, sex,severity) and progress (Experimental): the relation between progress in gross motor functions
  Interventions: Other: physical therapy intervention

INTERVENTIONS:
Other: physical therapy intervention — NDT bases on neuroplasticity by which the brain change and reorganize itself and its processes according to practice and experience by a) facilitation of normal postural alignment and movement patterns; b) inhibition of the involvement during developmental and functional activities; and c) using sensory feedback (manual contact, visual integration, somatosensory reinforcement) for recovering function
  Other Names: neurodevelopmental technique; strength training

SUMMARY:
The main outcome of physical therapy interventions is the progress of gross motor functions which result from the interactions between many factors not limited to physical, medical or surgical interventions but also including child characteristics and socializing agents. Aim of the study: To determine the effect of socioeconomic status (SES), child characteristics (age, sex, severity, and type of cerebral palsy) on the progress of gross motor functions in children with cerebral palsy. Methods: Prospective cohort study on eighty children (44 boys, 36 girls) aging 3.11 ± 0.88 years old, diagnosed as spastic cerebral palsy. The gross motor function measure (GMFM-88) between two-time intervals with follow-up time 6 months Results: The median of the mean difference for the GMFM scores was related to socioeconomic status, age, sex, severity, and type of CP.

DETAILED DESCRIPTION:
This study had four stages, the first one make registry from a computer database of outpatient clinic faculty of physical therapy Cairo university for all children with cerebral palsy under four years old age. In the second stage the files of 100 children registered were studied to select spastic cerebral palsy without the following; associated disorders, congenital anomalies, perceptual disorders, IQ below 80%, or another diagnosis ( nerve lesion, genetic disorders). Before the evaluation stage, every parent of each selected child was aware with the purpose of the study and signed the written informed consent that was approved by the ethical committee faculty of Physical Therapy Cairo University.Evaluation

The 83 selected children were evaluated as follow:

1. Muscle tone assessment Modified Ashworth scale is a valid and reliable test for measure muscle tone (Mutlu, 2008) table 1. Then evaluate the tone distribution throughout the body to determine its type diplegia, quadriplegia, or hemiplegia.
2. Severity The gross motor function classification system (GMFCS) is a reliable and valid system to classify the children with CP according to their age- specific motor activity (Palisano, 2000). GMFCS is a time-independent variable and it has five levels of severity (I, II, III, IV &V). The children with level I& II grouped as mild cases, children with level III were moderate cases, and those with IV & V levels were sever cases.
3. The gross motor function measure The Gross motor function measure (GMFM-88) is a valid clinical assessment tool designed to evaluate gross motor function, and its change over time in children with cerebral palsy (Russell, 2013). (GMFM-88) consists of 88 items in five dimensions A: Lying and Rolling (17 items), B: Sitting (20 items), C: Crawling and Kneeling (14 items), D: Standing (13 items), and E: Walking, Running and Jumping( 24 items). Each item was scored as 0 - does not initiate, 1 - initiates, 2 - partially completes, and 3 - completed, or not tested. The GMFM total scores are a summation of the scores for all dimensions and dividing by 5. A percentage score was calculated for the total score so it ranges from 0 to 100.
4. Socioeconomic status (SES) SES was evaluated by a valid and updated of the socioeconomic status scale for health research in Egypt scale (El-Gilany, 2012). It includes 7 domains with a total score of 84 ; 1- education and cultural domain(for both husband & wife) (score = 30); 2- family domain (score = 10); 3- occupation domain(for both husband & wife) (score = 10); 4- Family possessions domain (score = 12); 5- home sanitation domain (score = 12); 6- health care domain (score = 5); 7- economic domain(score = 5). According to the quartiles of the score calculated, the socioeconomic level is classified into very low, low, middle and high levels.

Physical therapy program The trained physiotherapists did the physical therapy interventions based on neurodevelopmental technique (NDT) and strength training for all participated children in the study for three times per week along sex months. During the study, the parents were asked to be adhering to the sessions Follow up After 6 months of the physical therapy program, the GMFM88 for 80 children were evaluated again to determine the progress of motor functions.

ELIGIBILITY:
Inclusion Criteria:

* all children with spastic cerebral palsy under four years old age

Exclusion Criteria:

* with associated disorders, congenital anomalies, perceptual disorders, had IQ below 80% or had another diagnosis ( nerve lesion, genetic disorders).

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
gross motor function measure | 20 minutes
  The Gross motor function measure (GMFM-88) is a valid clinical assessment tool designed to evaluate gross motor function, and its change over time in children with cerebral palsy (Russell, 2013). (GMFM-88) consists of 88 items in five dimensions A: Lying and Rolling (17 items), B: Sitting (20 items), C: Crawling and Kneeling (14 items), D: Standing (13 items), and E: Walking, Running and Jumping( 24 items). Each item was scored as 0 - does not initiate, 1 - initiates, 2 - partially completes, and 3 - completed, or not tested. The GMFM total scores is summation of the scores for all dimensions and dividing by 5. A percentage score was calculated for total score so it ranges from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: zeinab hussein, Principal Investigator — pediatric physical therapy
Locations (1):
- Zeinab Hussein, Cairo, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
on line publication
Supporting Information: Study Protocol
Time Frame: according to time of publication

REFERENCES:
- [Result] 1. Mutch L, Alberman E, Hagberg B, et al. Cerebral palsy epidemiology: where are we now and where are we going? Dev Med Child Neurol. 1992;34(6):547-51. [PubMed] [Google Scholar 2. Reeuwijk A, Van Schie PEM, Becher JG, et al. Effects of botulinum toxin type A on upper limb functions in children with cerebral palsy: a systematic review. Clin Rehabil. 2006;20(5):375-87. [PubMed] [Google Scholar]. 3. El-Tallawy, H. N., Farghaly, W. M., Shehata, G. A., Rageh, T. A., Metwally, N. A., Badry, R., … Kandil, M. R.. Cerebral palsy in Al-Quseir City, Egypt: prevalence, subtypes, and risk factors. Neuropsychiatric disease and treatment, 2014; 10, 1267-1272. 5- O'Shea TM, Preisser JS, Klinepeter KL, et al. Trends in mortality and cerebral palsy in a geographically based cohort of very low birth weight neonates born between1982 to 1994. Pediatrics. 1998;101(4 pt 1):642-[PubMed] [Google Scholar] 6- Shamsoddini AR, Hollisaz MT. Effect of sensory integration therapy on gross motor function in children with cerebral palsy. Iran J Child Neurology. 2009;3(1):43- 8. [Google Scholar] 7- McCullough N, Parkes J, Kerr C, McDowell BC(2013): The health of children and young people with cerebral palsy: a longitudinal, population-based study. Int J Nurs Stud. 50(6):747-756. [PubMed] [Google Scholar] 8- O'Shea, T. M. (2008). Diagnosis, treatment, and prevention of cerebral palsy in near-term/term infants. Clinical obstetrics and gynecology, 51(4), 816. 9- Saifi, S., & Mehmood, T. (2011). Effects of socio-economic status on students achievement. International Journal of Social Sciences and Education, 1(2), 119-128. 10- Braveman, P. A., Cubbin, C., Egerter, S., Chideya, S., Marchi, K. S., Metzler, M., & Posner, S. (2005). Socioeconomic status in health research: one size does not fit all. Jama, 294(22), 2879-2888. 11- Baker, E. H. (2014). Socioeconomic status, definition. The Wiley Blackwell Encyclopedia of health, illness, behavior, and society, 2210-2214. 12- Sundrum, R., Logan, S., Wallace, A., & Spencer, N. (2005). Cerebral palsy and socioeconomic status: a retrospective cohort study. Archives of disease in childhood, 90(1), 15-18. 13- Inchley, J. C., Currie, D. B., Todd, J. M., Akhtar, P. C., & Currie, C. E. (2005). Persistent socio-demographic differences in physical activity among Scottish schoolchildren 1990-2002. The European Journal of Public Health, 15(4), 386-388. 14- Myklebust G, Jahnsen R, Elkjaer S. (2009): Registration of interventions in children with cerebral palsy during three years-a population based study. [Scientific Poster Abstracts]. Developmental Medicine & Child Neurology. 51:65. doi: 10.1111/j.1469-8749.2009.03452_2.x 15- Palisano R, Begnoche DM, Chiarello LA, et al (2012): Amount and focus of physical therapy and occupational therapy for young children with cerebral palsy. Physical & occupational therapy in pediatrics. 32(4):368-82. doi: 10.3109/01942638.2012.715620. PubMed PMID: 22954372 16- Mutlu, A., Livanelioglu, A., & Gunel, M. K. (2008). Reliability of Ashworth and Modified Ashworth scales in children with spastic cerebral palsy. BMC musculoskeletal disorders, 9(1), 44. 17- Palisano, R. J., Hanna, S. E., Rosenbaum, P. L., Russell, D. J., Walter, S. D., Wood, E. P., ... & Galuppi, B. E. (2000). Validation of a model of gross motor function for children with cerebral palsy. Physical therapy, 80(10), 974-985. 18- WHO. (2001). International classification of functioning, disability and health: ICF. (World HealthOrganization. 19- Law,M., & Darrah, J. (2014). Emerging therapy approaches: An emphasis on function. Journal of ChildNeurology, 29(8), 1101-1107. doi:10.1177/0883073814533151 20- Anttila, H., Autti-Rämö, I., Suoranta, J., Mäkelä, M., & Malmivaara, A. (2008). Effectiveness of physical therapy interventions for children with cerebral palsy: a systematic review. BMC pediatrics, 8(1), 14. 21- Russell, D. J., Rosenbaum, P. L., Wright, M., & Avery, L. M. (2013). Gross Motor Function Measure (GMFM-66 & GMFM-88) User's Manual. High Holborn, UK, Mac Keith Press. 22- El-Gilany, A., El-Wehady, A., & El-Wasify, M. (2012). Updating and validation of the socioeconomic status scale for health research in Egypt. Eastern Mediterranean Health Journal, 18(9). 23- Huitt, W., & Hummel, J. (2003). Piaget's theory of cognitive development. Educational psychology interactive, 3(2), 1-5. 24- Malik, F., & Marwaha, R. (2018). Development, Stages of Social Emotional Development In Children. In StatPearls [Internet]. StatPearls Publishing.
- See also: selection of children — https://www.ncbi.nlm.nih.gov/books/NBK534819/
- Available data/document: Study Protocol — https://www.ncbi.nlm.nih.gov/